CLINICAL TRIAL: NCT06589804
Title: Randomized Phase III Trial of Pembrolizumab vs. Pembrolizumab/Cetuximab in Recurrent or Metastatic Head and Neck Squamous Cell Carcinoma With Platinum Refractory Disease
Brief Title: Testing the Addition of Anti-Cancer Drug, Cetuximab, to Standard of Care Treatment (Pembrolizumab) for Returning or Spreading Head and Neck Cancer After Previous Treatment
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2024-07339; NCI-2024-07339 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); A092205 (Other: Alliance for Clinical Trials in Oncology); A092205 (Other: CTEP); U10CA180821 (NIH)
Record Dates: First submitted 2024-09-06; First posted 2024-09-19 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-12

CONDITIONS: Metastatic Head and Neck Squamous Cell Carcinoma; Metastatic Hypopharyngeal Squamous Cell Carcinoma; Metastatic Laryngeal Squamous Cell Carcinoma; Metastatic Oral Cavity Squamous Cell Carcinoma; Metastatic Oropharyngeal Squamous Cell Carcinoma; Recurrent Head and Neck Squamous Cell Carcinoma; Recurrent Hypopharyngeal Squamous Cell Carcinoma; Recurrent Laryngeal Squamous Cell Carcinoma; Recurrent Neck Squamous Cell Carcinoma of Unknown Primary; Recurrent Oral Cavity Squamous Cell Carcinoma; Recurrent Oropharyngeal Squamous Cell Carcinoma; Refractory Head and Neck Squamous Cell Carcinoma; Refractory Hypopharyngeal Squamous Cell Carcinoma; Refractory Laryngeal Squamous Cell Carcinoma; Refractory Oral Cavity Squamous Cell Carcinoma; Refractory Oropharyngeal Squamous Cell Carcinoma; Stage IV Head and Neck Cutaneous Squamous Cell Carcinoma AJCC v8; Stage IV Hypopharyngeal Carcinoma AJCC v8; Stage IV Laryngeal Cancer AJCC v8; Stage IV Lip and Oral Cavity Cancer AJCC v8; Stage IV Oropharyngeal (p16-Negative) Carcinoma AJCC v8
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Hypopharyngeal Neoplasms; Laryngeal Neoplasms; Mouth Neoplasms; Carcinoma | interventions — Specimen Handling; Cetuximab; (225)Ac-DOTA-c(RGDyK); Magnetic Resonance Spectroscopy; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1 (pembrolizumab) (Active Comparator): Patients receive pembrolizumab IV over 30 minutes on day 1 of each cycle. Cycles repeat every 42 days for up to 18 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo CT, PET/CT or MRI throughout the trial and optionally undergo blood sample collection on study and at disease progression or end of treatment.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Biological: Pembrolizumab; Procedure: Positron Emission Tomography
- Arm 2 (cetuximab, pembrolizumab) (Experimental): Patients receive cetuximab IV over 120 minutes on day -14 prior to cycle 1 and then on days 1, 15 and 29 of each cycle and pembrolizumab IV over 30 minutes on day 1 of each cycle. Cycles repeat every 42 days for up to 18 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo CT, PET/CT or MRI throughout the trial and optionally undergo blood sample collection on study and at disease progression or end of treatment.
  Interventions: Procedure: Biospecimen Collection; Biological: Cetuximab; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Biological: Pembrolizumab; Procedure: Positron Emission Tomography

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Biological: Cetuximab — Given IV
  Other Names: C 225; C-225; C225; Cetuximab Biosimilar CDP-1; Cetuximab Biosimilar CMAB009; Cetuximab Biosimilar KL 140; Chimeric Anti-EGFR Monoclonal Antibody; Chimeric MoAb C225; Chimeric Monoclonal Antibody C225; Erbitux; IMC-C225
  Arms: Arm 2 (cetuximab, pembrolizumab)
Procedure: Computed Tomography — Undergo CT or PET/CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Biological: Pembrolizumab — Given IV
  Other Names: BCD-201; GME 751; GME751; Keytruda; Lambrolizumab; MK 3475; MK-3475; MK3475; Pembrolizumab Biosimilar BCD-201; Pembrolizumab Biosimilar GME751; Pembrolizumab Biosimilar QL2107; Pembrolizumab Biosimilar RPH-075; Pembrolizumab Biosimilar SB27; QL2107; RPH 075; RPH-075; RPH075; SB 27; SB-27; SB27; SCH 900475; SCH-900475; SCH900475
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT

SUMMARY:
This phase III trial compares the effect of adding cetuximab to pembrolizumab versus pembrolizumab alone in treating patients with head and neck squamous cell carcinoma (HNSCC) that has come back after a period of improvement (recurrent) and/or that has spread from where it first started (primary site) to other places in the body (metastatic). Cetuximab is in a class of medications called monoclonal antibodies. It binds to a protein called EGFR, which is found on some types of tumor cells. This may help keep tumor cells from growing. Immunotherapy with monoclonal antibodies, such as pembrolizumab, may help the body's immune system attack the tumor, and may interfere with the ability of tumor cells to grow and spread. Giving cetuximab and pembrolizumab together may be more effective at treating patients with recurrent and/or metastatic HNSCC than pembrolizumab alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess whether the combination of cetuximab and pembrolizumab (arm 2) compared to pembrolizumab alone (arm 1) results in improved overall survival (OS) in subjects with platinum refractory HNSCC.

SECONDARY OBJECTIVES:

I. To compare pembrolizumab + cetuximab (arm 2) versus (vs.) pembrolizumab alone (arm 1) with respect to objective response rate per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.

II. To compare pembrolizumab + cetuximab (arm 2) vs. pembrolizumab alone (arm 1) with respect to progression free survival (PFS) per RECIST 1.1.

III. To evaluate pembrolizumab + cetuximab (arm 2) vs. pembrolizumab alone (arm 1) with respect to duration of response (DOR) per RECIST 1.1.

IV. To assess the safety and tolerability of pembrolizumab + cetuximab (arm 2) vs. pembrolizumab alone (arm 1).

V. To assess the patient-reported toxicity using Patient Reported Outcomes version of Common Terminology Criteria for Adverse Events (PRO-CTCAE) of pembrolizumab + cetuximab (arm 2) vs. pembrolizumab alone (arm 1).

EXPLORATORY OBJECTIVES:

I. To identify specific mutational changes that may be indicative of clinical response to pembrolizumab + cetuximab and pembrolizumab alone.

II. To evaluate circulating tumor-derived deoxyribonucleic acid (ctDNA) kinetics over the course of treatment in response to pembrolizumab + cetuximab and pembrolizumab alone.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM 1: Patients receive pembrolizumab intravenously (IV) over 30 minutes on day 1 of each cycle. Cycles repeat every 42 days for up to 18 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo computed tomography (CT), positron emission tomography (PET)/CT or magnetic resonance imaging (MRI) throughout the trial and optionally undergo blood sample collection on study and at disease progression or end of treatment.

ARM 2: Patients receive cetuximab IV over 120 minutes on day -14 prior to cycle 1 and then on days 1, 15 and 29 of each cycle and pembrolizumab IV over 30 minutes on day 1 of each cycle. Cycles repeat every 42 days for up to 18 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo CT, PET/CT or MRI throughout the trial and optionally undergo blood sample collection on study and at disease progression or end of treatment.

After completion of study treatment, patients are followed up within 4 weeks and then every 3 and/or 6 months for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis head and neck squamous cell carcinomas (HNSCC).
* Previously untreated for recurrent and/or metastatic disease incurable by local therapies.
* Primary tumor location of oral cavity, oropharynx, larynx, or hypopharynx.

  * Note: Other primary tumor sites of HNSCC, including nasopharynx primary tumor are not eligible. Unknown primary tumors may be eligible and can be enrolled at the discretion of the treatment team with approval by the study chair.
* Measurable disease.
* Must have platinum-refractory disease defined as disease progression during or ≤ 29 weeks after completion of definitive therapy (chemoradiation therapy) or adjuvant (post-operative) therapy.
* Patient must have a combined positive score PD-L1 positive (CPS >/= 1) tumor.
* Any radiation therapy must be completed >= 10 days prior to registration.
* Patients should not have received any prior treatment in the recurrent or metastatic setting.
* Prior therapy with neoadjuvant or induction anti PD-1/PD-L1 monoclonal antibody or cetuximab in the curative setting is allowed if last treatment dose was >= 26 weeks prior to registration without evidence of disease progression during that treatment period.
* Patient has not received a live vaccine within 30 days prior to registration.
* Patient does not have a history of any contraindication or has a severe hypersensitivity to any component of pembrolizumab or cetuximab (≥ grade 3).
* Patient has not received chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone or equivalent) or any other form of immunosuppressive therapy within 7 days prior to registration.
* Patient with oropharyngeal cancer only must have negative results from testing of human papillomavirus (HPV) status defined as p16 immunohistochemistry (IHC) and/or HPV in situ hybridization (ISH).

  * Note: A Clinical Laboratory Improvement Act (CLIA) certified circulating tumor HPV deoxyribonucleic acid (ctHPVDNA) assay can be used if tissue sample is not available.
* Age ≥ 18 years.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2.
* Absolute neutrophil count (ANC) ≥ 1,500/mm^3.
* Platelet count ≥ 100,000/mm^3.
* Hemoglobin (Hgb) ≥ 9 g/dL (if < 9 g/dL, then transfusions are acceptable to increase hemoglobin above 9 g/dL).
* Creatinine ≤ 1.5 x upper limit of normal (ULN) OR calculated (calc.) creatinine clearance ≥ 30 mL/min using the Cockcroft-Gault formula for participant with creatinine levels > 1.5 x institutional ULN.
* Total bilirubin ≤ 1.5 x ULN OR direct bilirubin < ULN for participant with total bilirubin > 1.5 x institutional ULN.
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamic-pyruvic transaminase [SGPT]) ≤ 3.0 x ULN unless liver metastases are present in which case < 5.0 x ULN.
* Not pregnant and not nursing, because this study involves an agent that has known genotoxic, mutagenic, and teratogenic effects.

  * Therefore, for women of childbearing potential only, a negative pregnancy test done ≤ 7 days prior to registration is required.
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen should be included.
* For treated/stable brain metastases: Patients with treated brain metastases are eligible if follow-up brain imaging after central nervous system (CNS)-directed therapy shows no evidence of progression.

  * Patients with new or progressive brain metastases (active brain metastases) or leptomeningeal disease are eligible if the treating physician determines that immediate CNS specific treatment is not required and is unlikely to be required during the first cycle of therapy.
* HIV-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months prior to registration are eligible for this trial.
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated.
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load.
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class 2B or better.
* Patients does not have a history of active myocarditis.
* Patients does not have a history of any form of pneumonitis or diffuse idiopathic or immune mediated interstitial pulmonary disease.
* Patient does not have a history of solid organ transplantation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Estimated)
Dates: Start 2025-03-27 (Actual); Primary Completion 2029-11-30 (Estimated); Study Completion 2029-11-30 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | Time from randomization to death from any cause, assessed up to 5 years
  Will be estimated using the Kaplan-Meier method. Will be based on the stratified log-rank test that will compare the distributions across the treatment arms. Univariable and multivariable Cox models stratified by the stratification factors used in the randomization will be assessed as well, where the multivariable Cox model will also adjust for other key baseline factors of interest. Hazard ratios and 95% confidence intervals, along with likelihood ratio p-values will be reported from these Cox models.

SECONDARY OUTCOMES:
Confirmed response rate | Up to 5 years
  Will be assessed per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria if patients have a partial or complete response for 2 consecutive evaluations at least 4 weeks apart, using local review only. The proportion of patients with a confirmed response will be calculated and compared between the 2 arms using a Chi-square or Fisher's Exact test.
Duration of response | From the date at which the patient's earliest best objective status is first noted to be either a complete response or partial response to the earliest date progression is documented, assessed up to 5 years
  Will be defined for all evaluable patients who have achieved an objective response. Will be assessed per RECIST 1.1 criteria. Will be compared between the 2 arms using the Kaplan-Meier method, where the log-rank test will be used to compare the 2 treatment arms.
Progression free survival | Time from randomization to the first of either disease progression or death from any cause, assessed up to 5 years
  Disease progression will be assessed per RECIST 1.1 criteria. Will be compared between the 2 arms using the Kaplan-Meier method, where the log-rank test will be used to calculate the p-value.
Incidence of adverse events | Up to 5 years
  Will be summarized using Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. The frequency and percentage of grade 3+ adverse events will be compared between the 2 treatment arms. Comparisons between arms will be made by using either the Chi-square or Fisher's Exact test.
Patient-reported toxicity | Up to 5 years
  Will be assessed using Patient-Reported Outcomes version of the CTCAE. The frequency and proportion of patients with a maximum post-baseline score greater than 0 will be compared across arms using a Chi-square or Fisher's exact test with a nominal significance level of alpha = 0.10. Similarly, the frequency and proportion of patients with a maximum post-baseline score greater than or equal to 3 will be compared across arms using a Chi-square or Fisher's exact test with a nominal significance level of alpha = 0.10. Patients' maximum baseline-adjusted scores will be calculated using the method described by Dueck et al.

OTHER OUTCOMES:
Estimates of median OS by sex | Up to 5 years
  Estimates of treatment effects (median OS) and the corresponding 95% confidence intervals will be provided by sex.
Estimates of median OS by race | Up to 5 years
  Estimates of treatment effects (median OS) and the corresponding 95% confidence intervals will be provided by race.
Estimates of median OS by ethnicity | Up to 5 years
  Estimates of treatment effects (median OS) and the corresponding 95% confidence intervals will be provided by ethnicity.

CONTACTS AND LOCATIONS:
Overall Officials: Siddharth Sheth, Principal Investigator — Alliance for Clinical Trials in Oncology
Locations (172):
- United States (172):
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Fremont - Rideout Cancer Center, Marysville, California
  - VA Palo Alto Health Care System, Palo Alto, California
  - UCHealth Memorial Hospital Central, Colorado Springs, Colorado
  - Memorial Hospital North, Colorado Springs, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Cancer Care and Hematology-Fort Collins, Fort Collins, Colorado
  - Lutheran Hospital - Cancer Centers of Colorado, Golden, Colorado
  - UCHealth Greeley Hospital, Greeley, Colorado
  - Medical Center of the Rockies, Loveland, Colorado
  - Mount Sinai Medical Center, Miami Beach, Florida
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Clinic Cancer Services - Sandpoint, Sandpoint, Idaho
  - Advocate Good Shepherd Hospital, Barrington, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Advocate Illinois Masonic Medical Center, Chicago, Illinois
  - AMG Crystal Lake - Oncology, Crystal Lake, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Advocate Good Samaritan Hospital, Downers Grove, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Advocate Sherman Hospital, Elgin, Illinois
  - Advocate South Suburban Hospital, Hazel Crest, Illinois
  - AMG Libertyville - Oncology, Libertyville, Illinois
  - Condell Memorial Hospital, Libertyville, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - UC Comprehensive Cancer Center at Silver Cross, New Lenox, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Advocate Outpatient Center - Oak Lawn, Oak Lawn, Illinois
  - University of Chicago Medicine-Orland Park, Orland Park, Illinois
  - Advocate High Tech Medical Park, Palos Heights, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - UW Health Carbone Cancer Center Rockford, Rockford, Illinois
  - Memorial Hospital East, Shiloh, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - UChicago Medicine Northwest Indiana, Crown Point, Indiana
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic - Ames, Ames, Iowa
  - McFarland Clinic - Boone, Boone, Iowa
  - Mercy Hospital, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - McFarland Clinic - Trinity Cancer Center, Fort Dodge, Iowa
  - McFarland Clinic - Jefferson, Jefferson, Iowa
  - McFarland Clinic - Marshalltown, Marshalltown, Iowa
  - HaysMed, Hays, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - The University of Kansas Cancer Center - Olathe, Olathe, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - University of Kansas Hospital-Indian Creek Campus, Overland Park, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - University of Kansas Health System Saint Francis Campus, Topeka, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Brighton, Brighton, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Canton, Canton, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Chelsea Hospital, Chelsea, Michigan
  - Cancer Hematology Centers - Flint, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology Ann Arbor Campus, Ypsilanti, Michigan
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - University Health Truman Medical Center, Kansas City, Missouri
  - University of Kansas Cancer Center - Briarcliff, Kansas City, Missouri
  - University of Kansas Cancer Center - North, Kansas City, Missouri
  - University of Kansas Cancer Center - Lee's Summit, Lee's Summit, Missouri
  - Lake Regional Hospital, Osage Beach, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Jefferson Cherry Hill Hospital, Cherry Hill, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Sidney Kimmel Cancer Center Washington Township, Sewell, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Glens Falls Hospital, Glens Falls, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - SUNY Upstate Medical Center-Community Campus, Syracuse, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - Upstate Cancer Center at Verona, Verona, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Margaret R Pardee Memorial Hospital, Hendersonville, North Carolina
  - FirstHealth of the Carolinas-Moore Regional Hospital, Pinehurst, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Miami Valley Hospital South, Centerville, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Miami Valley Cancer Care and Infusion, Greenville, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Cancer Centers of Southwest Oklahoma Research, Lawton, Oklahoma
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Saint Alphonsus Cancer Care Center-Ontario, Ontario, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Pocono Medical Center, East Stroudsburg, Pennsylvania
  - Jefferson Torresdale Hospital, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Avera Cancer Institute - Mitchell, Mitchell, South Dakota
  - Avera Cancer Institute at Pierre, Pierre, South Dakota
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Avera Cancer Institute at Yankton, Yankton, South Dakota
  - VCU Massey Cancer Center at Stony Point, Richmond, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - West Virginia University Charleston Division, Charleston, West Virginia
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Aurora Saint Luke's South Shore, Cudahy, Wisconsin
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - ProHealth D N Greenwald Center, Mukwonago, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - ProHealth Waukesha Memorial Hospital, Waukesha, Wisconsin
  - UW Cancer Center at ProHealth Care, Waukesha, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm